CLINICAL TRIAL: NCT02817087
Title: An Innovative Approach to Restoration of Function in Chronic Ischemic Stroke Using a New Wearable Multifocal Brain Stimulator
Brief Title: Multifocal Brain Magnetic Stimulation in Chronic Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Chiu, MD (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Seraya Medical (Industry)
Responsible Party: Sponsor-Investigator, David Chiu, MD, Principal Investigator/Sponsor-Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00014213
Record Dates: First submitted 2016-03-31; First posted 2016-06-29 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Stroke
Keywords: Stroke; chronic ischemic stroke; cerebrovascular accident (CVA); ischaemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Transcranial Magnetic Stimulation; Control Groups

STUDY DESIGN:
Intervention Model Description: Active repetitive transcranial magnetic stimulation administered through cap worn by patient under healthcare provider.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind, only the care provider is aware of active treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- repetitive Transcranial Magnetic Stimulation -On (Active Comparator): Participants wear the repetitive transcranial magnetic stimulation (rTMS) cap delivering magnetic stimulation to part of the brain.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation -On
- repetitive Transcranial Magnetic Stimulation -Off (Sham Comparator): Participants wear the repetitive transcranial magnetic stimulation (rTMS) cap that does NOT delivery any magnetic stimulation to the brain.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation -Off

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation -On — Cap worn on the scalp will deliver active Repetitive Transcranial Magnetic Stimulation to specific parts of the brain
  Other Names: transcranial magnetic stimulation (TMS); Transcranial Rotating Permanent Magnet Stimulation (TRPMS); repetitive Transcranial Magnetic Stimulation (rTMS)
  Arms: repetitive Transcranial Magnetic Stimulation -On
Device: repetitive Transcranial Magnetic Stimulation -Off — Cap worn on the scalp will no delivery of the Repetitive Transcranial Magnetic Stimulation to any part of the, referred to as a sham or inactive study treatment.
  Other Names: sham treatment; Control Group
  Arms: repetitive Transcranial Magnetic Stimulation -Off

SUMMARY:
Transcranial magnetic stimulation for post-stroke upper-body motor deficits.

DETAILED DESCRIPTION:
This study uses transcranial magnetic stimulation (magnetic pulses delivered through a specially designed cap worn on the head aimed at specific motor areas of the brain (brain areas responsible for the body's physical movements) to test whether upper-body motor function can be improved.

This is a double-blind study where half of participants will receive active transcranial stimulation and the other half of the participants will receive no transcranial magnetic stimulation; all participants will wear the cap. Participants and some members of the research team will not know who received active magnetic brain stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years;
* Clinical diagnosis of chronic ischemic stroke recovering for more than 3 months with unilateral motor deficits of arm and leg, or arm alone; --

Exclusion Criteria:

* History of seizure;
* Epileptogenic activity (indicative of increased risk of seizures) on EEG;
* Any active unstable medical condition;
* Pregnancy;
* Schizophrenia, bipolar disorder, alcoholism, or substance abuse;
* Medications which in the investigator's clinical judgment significantly lower the seizure threshold;
* Presence of metal or electronic implants in the head (or any in the body that preclude MRI) , including pacemakers, defibrillators, aneurysm clips, neuro-stimulators, cochlear implants, metal in the eyes, etc.;
* Any changes in medications prescribed for the treatment of stroke impairment within six weeks prior to inclusion in the study or at any time during the study.
* Botulinum toxin use within two months prior to the screening visit or any planned use of botulinum toxin during the study
* Changes in NIHSS and motor assessment scores between Visit 1 and Visit 2 indicating that the patient's impairment is not stable. The following cutoffs, based on research establishing Clinically Important Differences, will be used for this determination:
* National Institutes of Health Stroke Scale: A change in total score of more than 2 points in either direction, or a change in the motor extremity score of more than 1 point in either direction.
* Fugl-Meyer Assessment of Sensorimotor Impairment: A change of more than 5 points in either direction on the upper-extremity motor score for the affected arm.
* Action Research Arm Test: A change of more than 5 points in either direction on the ARAT score for the affected arm.
* Any condition that precludes a high quality brain MRI scan.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Chiu, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rehme AK, Grefkes C. Cerebral network disorders after stroke: evidence from imaging-based connectivity analyses of active and resting brain states in humans. J Physiol. 2013 Jan 1;591(1):17-31. doi: 10.1113/jphysiol.2012.243469. Epub 2012 Oct 22. PMID 23090951
- [Background] Li W, Li Y, Zhu W, Chen X. Changes in brain functional network connectivity after stroke. Neural Regen Res. 2014 Jan 1;9(1):51-60. doi: 10.4103/1673-5374.125330. PMID 25206743
- [Background] Varsou O, Macleod MJ, Schwarzbauer C. Functional connectivity magnetic resonance imaging in stroke: an evidence-based clinical review. Int J Stroke. 2014 Feb;9(2):191-8. doi: 10.1111/ijs.12033. Epub 2013 Mar 19. PMID 23506092
- [Background] Ameli M, Grefkes C, Kemper F, Riegg FP, Rehme AK, Karbe H, Fink GR, Nowak DA. Differential effects of high-frequency repetitive transcranial magnetic stimulation over ipsilesional primary motor cortex in cortical and subcortical middle cerebral artery stroke. Ann Neurol. 2009 Sep;66(3):298-309. doi: 10.1002/ana.21725. PMID 19798637
- [Background] Chang WH, Kim YH, Bang OY, Kim ST, Park YH, Lee PK. Long-term effects of rTMS on motor recovery in patients after subacute stroke. J Rehabil Med. 2010 Sep;42(8):758-64. doi: 10.2340/16501977-0590. PMID 20809058
- [Background] Kim YH, You SH, Ko MH, Park JW, Lee KH, Jang SH, Yoo WK, Hallett M. Repetitive transcranial magnetic stimulation-induced corticomotor excitability and associated motor skill acquisition in chronic stroke. Stroke. 2006 Jun;37(6):1471-6. doi: 10.1161/01.STR.0000221233.55497.51. Epub 2006 May 4. PMID 16675743
- [Background] Khedr EM, Etraby AE, Hemeda M, Nasef AM, Razek AA. Long-term effect of repetitive transcranial magnetic stimulation on motor function recovery after acute ischemic stroke. Acta Neurol Scand. 2010 Jan;121(1):30-7. doi: 10.1111/j.1600-0404.2009.01195.x. Epub 2009 Aug 11. PMID 19678808
- [Background] Fitzgerald PB, Fountain S, Daskalakis ZJ. A comprehensive review of the effects of rTMS on motor cortical excitability and inhibition. Clin Neurophysiol. 2006 Dec;117(12):2584-96. doi: 10.1016/j.clinph.2006.06.712. Epub 2006 Aug 4. PMID 16890483
- [Background] Fregni F, Boggio PS, Valle AC, Rocha RR, Duarte J, Ferreira MJ, Wagner T, Fecteau S, Rigonatti SP, Riberto M, Freedman SD, Pascual-Leone A. A sham-controlled trial of a 5-day course of repetitive transcranial magnetic stimulation of the unaffected hemisphere in stroke patients. Stroke. 2006 Aug;37(8):2115-22. doi: 10.1161/01.STR.0000231390.58967.6b. Epub 2006 Jun 29. PMID 16809569
- [Background] Mally J, Dinya E. Recovery of motor disability and spasticity in post-stroke after repetitive transcranial magnetic stimulation (rTMS). Brain Res Bull. 2008 Jul 1;76(4):388-95. doi: 10.1016/j.brainresbull.2007.11.019. Epub 2007 Dec 26. PMID 18502315
- [Background] Boggio PS, Alonso-Alonso M, Mansur CG, Rigonatti SP, Schlaug G, Pascual-Leone A, Fregni F. Hand function improvement with low-frequency repetitive transcranial magnetic stimulation of the unaffected hemisphere in a severe case of stroke. Am J Phys Med Rehabil. 2006 Nov;85(11):927-30. doi: 10.1097/01.phm.0000242635.88129.38. PMID 17079967
- [Background] Grefkes C, Nowak DA, Wang LE, Dafotakis M, Eickhoff SB, Fink GR. Modulating cortical connectivity in stroke patients by rTMS assessed with fMRI and dynamic causal modeling. Neuroimage. 2010 Mar;50(1):233-42. doi: 10.1016/j.neuroimage.2009.12.029. Epub 2009 Dec 18. PMID 20005962
- [Background] Helekar, S.A., et al., Electromyographic motor-evoked potentials elicited by transcranial magnetic stimulation with rapidly moving permanent magnets mounted on a multisite stimulator cap, in 2013 Neuroscience Meeting Planner. 2013, Society for Neuroscience: San Diego, CA.
- [Background] Ashburner J, Friston KJ. Nonlinear spatial normalization using basis functions. Hum Brain Mapp. 1999;7(4):254-66. doi: 10.1002/(SICI)1097-0193(1999)7:4<254::AID-HBM4>3.0.CO;2-G. PMID 10408769
- [Background] Tzourio-Mazoyer N, Landeau B, Papathanassiou D, Crivello F, Etard O, Delcroix N, Mazoyer B, Joliot M. Automated anatomical labeling of activations in SPM using a macroscopic anatomical parcellation of the MNI MRI single-subject brain. Neuroimage. 2002 Jan;15(1):273-89. doi: 10.1006/nimg.2001.0978. PMID 11771995
- [Background] Bressler SL, Seth AK. Wiener-Granger causality: a well established methodology. Neuroimage. 2011 Sep 15;58(2):323-9. doi: 10.1016/j.neuroimage.2010.02.059. Epub 2010 Mar 2. PMID 20202481
- [Background] Matias FS, Gollo LL, Carelli PV, Bressler SL, Copelli M, Mirasso CR. Modeling positive Granger causality and negative phase lag between cortical areas. Neuroimage. 2014 Oct 1;99:411-8. doi: 10.1016/j.neuroimage.2014.05.063. Epub 2014 Jun 2. PMID 24893321
- [Background] Chen Y, Bressler SL, Ding M. Frequency decomposition of conditional Granger causality and application to multivariate neural field potential data. J Neurosci Methods. 2006 Jan 30;150(2):228-37. doi: 10.1016/j.jneumeth.2005.06.011. Epub 2005 Aug 15. PMID 16099512
- [Background] Blair RC, Karniski W. An alternative method for significance testing of waveform difference potentials. Psychophysiology. 1993 Sep;30(5):518-24. doi: 10.1111/j.1469-8986.1993.tb02075.x. PMID 8416078
- [Background] Chiavarini M, Morini G, Barocelli E, Bordi F, Plazzi PV, Vitali T, Impicciatore M. Influence of urea-equivalent groups in position 5 of 2-amino, 2-(1-aminoethylidenamino) and 2-guanidino thiazole derivatives on H2-receptor antagonist activity in gastric fistula cat. Agents Actions. 1989 Apr;27(1-2):192-4. doi: 10.1007/BF02222236. PMID 2568739
- [Background] Carlowe J. Investigation into home care of elderly people shows cases of "serious neglect". BMJ. 2011 Jun 21;342:d3904. doi: 10.1136/bmj.d3904. No abstract available. PMID 21693536
- [Background] S. A. Helekar and H. U. Voss,

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 patients were screened 7 were screen fails. 2 withdrawn. 14 treated-Active, 15 treated-placebo.
Period: Overall Study
Arm/Group | Repetitive Transcranial Magnetic Stimulation -On | Repetitive Transcranial Magnetic Stimulation -Off
Started | 16 | 15
Completed | 14 (1 pt was withdrawn early d/t concurrent disease. One pt. withdrew ICF d/t transportation concerns) | 15
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: 1 pt was withdrawn early d/t concurrent disease. One pt. withdrew ICF d/t transportation concerns
Groups:
- Total: Total of all reporting groups
Arm/Group | Repetitive Transcranial Magnetic Stimulation -On | Repetitive Transcranial Magnetic Stimulation -Off | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants] — Population: 1 pt was withdrawn early d/t concurrent disease. One pt. withdrew ICF d/t transportation concerns
  Participants
    number analyzed (Participants) | 14 | 15 | 29
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 6 | 7 | 13
    >=65 years | 8 | 8 | 16
Age, Continuous [Mean (Full Range); unit: years] — Population: 1 pt was withdrawn early d/t concurrent disease. One pt. withdrew ICF d/t transportation concerns
  years
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 65.4 [47 to 78] | 66.3 [45 to 80] | 65.8 [45 to 80]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 pt was withdrawn early d/t concurrent disease. One pt. withdrew ICF d/t transportation concerns
  Participants
    number analyzed (Participants) | 14 | 15 | 29
    Female | 6 | 9 | 15
    Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: pt was withdrawn early d/t concurrent disease. One pt. withdrew ICF d/t transportation concerns
  Participants
    number analyzed (Participants) | 14 | 15 | 29
    Hispanic or Latino | 2 | 1 | 3
    Not Hispanic or Latino | 12 | 14 | 26
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: pt was withdrawn early d/t concurrent disease. One pt. withdrew ICF d/t transportation concerns
  Participants
    number analyzed (Participants) | 14 | 15 | 29
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 3 | 0 | 3
    White | 10 | 15 | 25
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: 1 pt was withdrawn early d/t concurrent disease. One pt. withdrew ICF d/t transportation concerns
  participants
    United States: number analyzed (Participants) | 14 | 15 | 29
    United States | 14 | 15 | 29
Fugl-Meyer motor arm score [Median (Inter-Quartile Range); unit: score on a scale] — Scale range is 0-66 with higher score representing a better outcome. Population: 1 pt was withdrawn early d/t concurrent disease. One pt. withdrew ICF d/t transportation concerns
  score on a scale
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 43 [16 to 56] | 25 [15 to 52] | 37.0 [15.75 to 54.25]
National Institutes of Health Stroke Scale (NIHSS) [Median (Inter-Quartile Range); unit: score on a scale] — Total score is 0-42, with the lower score representing a better outcome Population: 1 pt was withdrawn early d/t concurrent disease. One pt. withdrew ICF d/t transportation concerns
  score on a scale
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 3 [2 to 6] | 3 [1 to 5] | 3.0 [1.75 to 5.0]
Action Research Arm Test (ARAT) [Median (Inter-Quartile Range); unit: score on a scale] — Total score is 0-57 with the higher score representing a better outcome Population: 1 pt was withdrawn early d/t concurrent disease. One pt. withdrew ICF d/t transportation concerns
  score on a scale
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 29 [0 to 57] | 6 [0 to 53] | 14.0 [0.0 to 56.0]
Hand Grip Strength [Median (Inter-Quartile Range); unit: Pounds] — Population: 1 pt was withdrawn early d/t concurrent disease. One pt. withdrew ICF d/t transportation concerns
  Pounds
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 19.7 [0 to 44] | 30.6 [0 to 54.4] | 21.8 [0.0 to 46.48]
Pinch Strength [Median (Inter-Quartile Range); unit: Pounds] — Population: 1 pt was withdrawn early d/t concurrent disease. One pt. withdrew ICF d/t transportation concerns
  Pounds
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 6.5 [0 to 10] | 3.83 [1 to 9.67] | 4.7 [0.75 to 9.78]
Gait velocity on Timed Up and Go Test [Median (Inter-Quartile Range); unit: feet per second] — Population: 1 pt was withdrawn early d/t concurrent disease. One pt. withdrew ICF d/t transportation concerns
  feet per second
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 1.32 [0 to 1.69] | 1.45 [0 to 1.74] | 1.45 [0.0 to 1.7]

OUTCOME MEASURES:

1. Primary Outcome: Changes in Brain Activation
Description: Change in number of active voxels in the cortical areas surrounding the lesion on functional MRI
Time Frame: One business day before treatment begins, one business day after treatment ends, up to 5 weeks
Measure: Median (Inter-Quartile Range); unit: voxels
Arm/Group | Repetitive Transcranial Magnetic Stimulation -On | Repetitive Transcranial Magnetic Stimulation -Off
Number analyzed (Participants) | 14 | 15
voxels | 48.5 [-60 to 81] | -30 [-373.3 to 0]

2. Secondary Outcome: Fugl-Meyer Motor Arm Score
Description: Change in arm motor function Total score range is 0-66 with the higher number representing a better outcome
Time Frame: One business day before treatment begins, one business day after treatment ends up to 5 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Repetitive Transcranial Magnetic Stimulation -On | Repetitive Transcranial Magnetic Stimulation -Off
Number analyzed (Participants) | 14 | 15
score on a scale | 2.5 [0 to 6.0] | 2.0 [-1.0 to 8.0]

3. Secondary Outcome: ARAT (Action Research Arm Test)
Description: Change in arm and hand motor function Total score range is 0-57 with the higher number representing a better outcome
Time Frame: One business day before treatment begins, one business day after treatment ends up to 5 weeks
Population: Stroke patients greater than 3 months from qualifying stroke date
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Repetitive Transcranial Magnetic Stimulation -On | Repetitive Transcranial Magnetic Stimulation -Off
Number analyzed (Participants) | 14 | 15
score on a scale | 0 [0 to 3.0] | 0 [0 to 4.0]

4. Secondary Outcome: Hand Dynamometer
Description: Change in grip strength The higher the number represents better outcome
Time Frame: One business day before treatment begins, one business day after treatment ends up to 5 weeks
Measure: Median (Inter-Quartile Range); unit: pounds
Arm/Group | Repetitive Transcranial Magnetic Stimulation -On | Repetitive Transcranial Magnetic Stimulation -Off
Number analyzed (Participants) | 14 | 15
pounds | 1.8 [0 to 4.9] | 0 [-2.2 to 2.2]

5. Secondary Outcome: Pinch Dynamometer Score
Description: Change in pinch strength. The higher the number, the better the outcome.
Time Frame: One business day before treatment begins, one business day after treatment ends up to 5 weeks
Measure: Median (Inter-Quartile Range); unit: pounds
Arm/Group | Repetitive Transcranial Magnetic Stimulation -On | Repetitive Transcranial Magnetic Stimulation -Off
Number analyzed (Participants) | 14 | 15
pounds | .17 [0 to .67] | .33 [0 to .83]

6. Secondary Outcome: TUG (Timed Up and Go Test)
Description: Change in gait velocity on Timed Up and Go Test. The lower the time recorded, the better the outcome.
Time Frame: One business day before treatment begins, one business day after treatment ends up to 5 weeks
Measure: Median (Inter-Quartile Range); unit: feet per second
Arm/Group | Repetitive Transcranial Magnetic Stimulation -On | Repetitive Transcranial Magnetic Stimulation -Off
Number analyzed (Participants) | 14 | 15
feet per second | .04 [0 to .11] | 0 [-.11 to .12]

7. Secondary Outcome: National Institutes of Health Stroke Scale (NIHSS)
Description: Change in National Institutes of Health Stroke Scale (NIHSS) Total score range is 0-42 with the lower number representing a better outcome
Time Frame: One business day before treatment begins, one business day after treatment ends up to 5 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Repetitive Transcranial Magnetic Stimulation -On | Repetitive Transcranial Magnetic Stimulation -Off
Number analyzed (Participants) | 14 | 15
score on a scale | 0 [-1 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events were captured from time of first treatment to completion of the final visit at 3 months post treatment. Serious adverse events were captured from time of informed consent to completion of the final visit at 3 months post treatment.
Description: All reported events were assessed by the Principal Investigator and resulted in no withdrawals due to study treatment
Arm/Group | Repetitive Transcranial Magnetic Stimulation -On | Repetitive Transcranial Magnetic Stimulation -Off
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/16 | 2/15
Other Adverse Events (participants affected / at risk) | 1/16 | 3/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Repetitive Transcranial Magnetic Stimulation -On (N=16) | Repetitive Transcranial Magnetic Stimulation -Off (N=15)
Acute Ischemic Stroke (Nervous system disorders) | 1 (1) | 0 (0) — Relationship= Unlikely
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) — Relationship= Unlikely
Migraine (Nervous system disorders) | 0 (0) | 1 (1) — Relationship=Unlikely
Renal stone (Renal and urinary disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) — 3 weeks post-treatment. Relationship=Unlikely
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Repetitive Transcranial Magnetic Stimulation -On (N=16) | Repetitive Transcranial Magnetic Stimulation -Off (N=15)
Fall (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Muscle cramps (General disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 1 (1) | 1 (1)
Transient tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT02817087/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT02817087/ICF_001.pdf